CLINICAL TRIAL: NCT03959644
Title: Failure Rate in Spinal Blocks and Determination of Related Factors: A Cross-Sectional, Prospective, Observational Study
Brief Title: Failure Rate in Spinal Blocks and Determination of Related Factors
Status: Completed | Type: Observational
Sponsor: Bozyaka Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Afife Aysun Kar, Principal Investigator, Bozyaka Training and Research Hospital
Other Study IDs: Failure of Spinal Anesthesia
Record Dates: First submitted 2019-05-16; First posted 2019-05-22 (Actual); Last update posted 2022-10-25 (Actual); Status verified 2022-10

CONDITIONS: Anesthesia, Spinal
Keywords: unsuccessful spinal anesthesia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Investigators aimed to determine the rates of unsuccessful spinal anesthesia, to determine the factors related to failure and to determine the measures that may be taken to reduce this problem.

DETAILED DESCRIPTION:
The study is as a cross-sectional, prospective, observational. After institutional review board approval and informed written consent, all patients aged ≥ 18 years undergoing spinal anesthesia in the Izmir Bozyaka Training and Research Hospital Operating Room will be included in the study. The specialist and assistant physician in charge of spinal anesthesia management of patients will undertake their own routine anesthesia management and the researcher will not be involved in any way. Patients who underwent combined spinal-epidural anesthesia and patients without consent were excluded. The primary aim of the study was to determine the rate of unsuccessful spinal anesthesia (total failure and partial failure) and to determine the factors that may be associated with these. Total failure was described as failure of localization of subarachnoid space with lumbar puncture; no motor and / or sensory block occurring within 10 minutes after the injection of local anesthetic into the subarachnoid space; repeated spinal anesthesia or general anesthesia. Partial failure was described as the need for anesthetic agents such as ketamine, propofol or opioid for the intraoperative pain relief, except for the use of midazolam and fentanyl in order to increase the patient's comfort.The secondary aim of the study was to determine the first attempt success and related factors. The first attempt success was described as identification or subarachnoid space at the first attempt.

Parameters to be recorded during the study are: age, gender, weight, height, body mass index (BMI), American Society of Anesthesiologist (ASA) status, type of surgery, elective / emergency surgery, patient's body type, spinal anatomy, position of the patient and the practitioner during spinal intervention, the technique applied (median /paramedian), the level of puncture, the type of spinal needle, the direction of the spinal needle notch, the number of spinal puncture, the nature of the cerebrospinal fluid (CSF) (clear/haemorrhagic), whether or not aspiration is performed, whether or not free CSF is controlled before or after drug injection, whether the practitioner is an expert or assistant, the assistant is seniority year, the type of local anesthetic, if the adjuvant drug is added to the local anesthetic, the dose of anesthetic, the loss of drug during injection of local anesthesia, position of the patient after injection, duration of surgery, testing of motor and sensory block, what is done in case of unsuccessful spinal anesthesia, examination of sacral dermatomes prior to second spinal anesthesia intervention will be recorded. Parameters will be recorded by Anesthesia Specialist, Anesthesia Assistant or Anesthesia Technician. At the end of the case, the registration form will be left at the designated place in the Anesthesia Clinic room.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged ≥ 18 years who are undergoing spinal anesthesia in Izmir Bozyaka Training and Research Hospital during study period.
2. American Society of Anesthesiologist Physical Status classification (ASA) I-IV.

Exclusion Criteria:

1. Patients who are undergoing combined spinal-epidural anesthesia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients aged ≥ 18 years undergoing spinal anesthesia in the Izmir Bozyaka Training and Research Hospital Operating Room will be included in the study.
Sampling Method: Probability Sample
Enrollment: 1431 (Actual)
Dates: Start 2019-05-10 (Actual); Primary Completion 2020-05-10 (Actual); Study Completion 2020-05-10 (Actual)

PRIMARY OUTCOMES:
Determination of Total Failure | During spinal punction procedure
  1. Failure of localization of subarachnoid space with lumbar puncture and conversion from spinal anesthesia to general anesthesia
Determination of Total Failure | At 10 min after spinal anesthetic injection
  2. No motor block (Bromage Scale = 0) occurring within 10 minutes after the injection of local anesthetic into the subarachnoid space and performing spinal anesthesia for the second time or conversion from spinal anesthesia to general anesthesia.
  Motor block will be determined by Bromage scale. Bromage Scale: 0 = ability to lift an extended knee at the hip; 1 = ability to flex the knee but not to lift an extended leg; 2 = ability to flex toes only; 3 = inability to move.
Determination of Total Failure | At 10 min after spinal anesthetic injection
  No sensory block (Pinprick Test = 0) occurring within 10 minutes after the injection of local anesthetic into the subarachnoid space and performing spinal anesthesia for the second time or conversion from spinal anesthesia to general anesthesia.
  Sensory block will be determined by Pinprick test. Pinprick Test: Sensory 0 = an ability to appreciate a pinprick as sharp; 1 = perception of a pinprick as less sharp than in unblocked areas; 2 = perception of a pinprick as touch but not sharp (analgesia); 3 = an inability to feel pinprick (anesthesia).
Determination of Partial Failure | From the spinal anesthetic injection to end of the surgery.
  After complete spinal anesthesia, the need for intravenous anesthetic agents such as ketamine, propofol, opioid or general anesthesia in the intraoperative period for pain relief when a patient complained of moderate to severe pain or had a Visual Analogue Scale (VAS) of > 3 out of 10 from the surgical site.
  Visual Analogue Scale (VAS): 0 = No pain - 10 = Worst imaginable pain.

SECONDARY OUTCOMES:
The first attempt success | Before the spinal anesthetic injection
  Identification of subarachnoid space at first spinal puncture.

CONTACTS AND LOCATIONS:
Overall Officials: Aysun Afife Kar, Uz. Dr., Principal Investigator — Aysun Afife Kar
Locations (1):
- Bozyaka Training and Research Hospital, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No